CLINICAL TRIAL: NCT00958087
Title: 18F-fluorodeoxyglucose Positron Emission Tomography Imaging in Cardiac Sarcoidosis Reveals Characteristic Heterogeneity of Tracer Uptake and the Disease Activity in Myocardium
Brief Title: Cardiac Sarcoidosis and FDG-PET
Status: Completed | Type: Observational
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Nobuhiro Tahara, M.D., PhD, Kurume University
Other Study IDs: CS-PET
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2010-07

CONDITIONS: Sarcoidosis; Dilated Cardiomyopathy
MeSH Terms: conditions — Sarcoidosis; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Sarcoidosis with cardiac involvement
- Dilated cardiomyopathy
- Sarcoidosis without cardiac involvement
- Healthy controls

SUMMARY:
Sarcoidosis is a multi-systemic inflammatory disorder of unknown cause characterized by the formation of non-caseating granulomas in involved organs. Its cardiac involvement may be potentially fatal. Although endomyocardial biopsy is required for deﬁnitive diagnosis of cardiac sarcoidosis, it is invasive and lacks sensitivity. The specific diagnostic tool for cardiac sarcoidosis is far from satisfactory. Recent studies have revealed that FDG-PET with under fasting conditions is a useful method for identiﬁcation of cardiac sarcoidosis patients. However, to our knowledge, no investigations have been published with regard to FDG quantification for the diagnosis and management of cardiac sarcoidosis by PET.

DETAILED DESCRIPTION:
Fasting FDG-PET will be performed in all subjects. Serum calcium, C-reactive protein (CRP), angiotensin converting enzyme (ACE), lysozyme, and B-type natriuretic peptide (BNP) levels will be measured in all patients. All patients will undergo chest X-ray, resting 12-lead ECG, transthoracic echocardiography, and 3 types of radionucleotide imaging using Tc-99m sestamibi for myocardial perfusion, Ga and FDG for whole-body evaluation. All assessments will be conducted within 2 weeks and no sign indicated any change in disease activity of sarcoidosis. The patients with cardiac involvement will be treated with 30 mg/day of prednisolone orally for the first 4 weeks, then will decrease to a dose of 20 mg/day for the next 4 weeks, and will maintain to a dose of 10 mg/day afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 35 and 85 years
* Subjects with systemic sarcoidosis
* Subjects with idiopathic sarcoidosis

Exclusion Criteria:

* Subjects with active inflammatory diseases not related to sarcoidosis
* Subjects with coronary artery disease and primary valvular heart diseases
* Subjects with uncontrolled diabetes mellitus or insulin treatment
* Subjects with use of the corticosteroid
* Subjects with systemic disorders such as active inflammatory, liver, renal, hematopoietic, and malignant disease

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fasting FDG-PET will be performed in patients with sarcoidosis and age-matched DCM patients. Among them, systemic sarcoidosis will be diagnosed clinically and/or histologically, and referred for cardiac sarcoidosis. Patients with sarcoidosis will reveal cardiac involvement based on guidelines established in 2006 by the Japanese Ministry of Health and Welfare. Healthy control subjects will undergo FDG-PET.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-03; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Usefulness of Fasting FDG-PET for Diagnosis and Management of Cardiac Sarcoidosis | Baseline and at 1, 3, 6, 12 months after the initial FDG-PET

SECONDARY OUTCOMES:
Change from baseline in circulating markers of inflammatory and sarcoidosis | Baseline and at 1, 3, 6, 12 months after the initial FDG-PET
Change from baseline in plasma dendritic cells | Baseline and at 1, 3, 6, 12 months after the initial FDG-PET
Change from baseline in plasma BNP, AGE, RAGE, and PEDF levels | Baseline and at 1, 3, 6, 12 months after the initial FDG-PET
All cardiovascular events and all cause death for 5 years | Baseline and at 1, 3, 6, 12 months after the initial FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhiro Tahara, MD, PhD, Principal Investigator — Kurume University
Locations (1):
- Kurume University Hospital, Kurume, Japan